CLINICAL TRIAL: NCT05977231
Title: Evaluation of Efficacy of Conservative Treatments in Women With Urinary Incontinence
Brief Title: Efficacy of Conservative Treatments for Urinary Incontinence in Women
Status: Recruiting | Type: Observational
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, The Office of Research and Development staff, Mackay Medical College
Other Study IDs: 23MMHIS058e
Record Dates: First submitted 2023-07-13; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Bladder training (BT): Data obtained before and after the training.
  Interventions: Procedure: BT
- biofeedback-assisted pelvic floor muscle training (bPFMT): Data obtained before and after the training.
  Interventions: Procedure: bPFMT
- intra-vaginal electric stimulation (iVES): Data obtained before and after the training.
  Interventions: Procedure: iVES
- BT+bPFMT: Data obtained before and after the training.
  Interventions: Procedure: BT + bPFMT
- BT+iVES: Data obtained before and after the training.
  Interventions: Procedure: BT + iVES
- bPFMT+iVES: Data obtained before and after the training.
  Interventions: Procedure: bPFMT + iVES

INTERVENTIONS:
Procedure: BT — A program of BT (including exercise and muscle training)
  Groups: Bladder training (BT)
Procedure: bPFMT — A bPFMT program at home
  Groups: biofeedback-assisted pelvic floor muscle training (bPFMT)
Procedure: iVES — An iVES program at home
  Groups: intra-vaginal electric stimulation (iVES)
Procedure: BT + bPFMT — Combination of BT and bPFMT
  Groups: BT+bPFMT
Procedure: BT + iVES — Combination of BT and iVES
  Groups: BT+iVES
Procedure: bPFMT + iVES — Combination of bPFMT and iVES
  Groups: bPFMT+iVES

SUMMARY:
To conduct a retrospective study to examine the effect of these conservative treatments to the symptoms and quality of life of patients with urinary incontinence. The investigators will use both subjective and objective assessment parameters, such as self-report symptoms, bladder diary, pad test and urodynamic study to access the improvement.

DETAILED DESCRIPTION:
Urinary incontinence is a common problem among women. The main types include stress incontinence, urge incontinence, and overflow incontinence. Other underlying pathology, such as cancer or neurologic disease can also cause urinary incontinence. To limit the medical expenses and possible complications of surgical treatment, the current treatment guidelines recommend conservative treatment as the first choice. According to American Urological Association (AUA)/Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction (SUFU) guidelines, the first-line treatment for non-neurologic overactive bladder should be behavioral therapy, such as bladder training, water restriction, and pelvic floor muscle training, physiological feedback, pessary, etc. Bladder training aims to increase the time interval between voids, and to increase the bladder capacity by self-adjusted schedules. Pelvic floor muscle training strengthens the pelvic floor muscles to provide urethral support to prevent urine leakage and suppress urgency. There is strong evidence that pelvic floor muscle training is beneficial for stress urinary incontinence.

The second-line treatment is medication, including anticholinergic drugs and ß3 adrenoceptor-acting agents. Anticholinergic drugs can reduce bladder detrusor contraction, and ß3 adrenoceptor-acting agents can relax the detrusor and increase bladder capacity.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patient diagnosed with urinary incontinence through clinical assessment
* Diagnosed at Mackay Memorial Hospital and underwent non-surgical treatment and subsequent follow-up.

Exclusion Criteria:

* Choosing invasive or surgical treatment options (such as bladder botulinum toxin injection, urethral sling surgery).
* Unable to comply with regular follow-up for at least one year.
* Pregnant women
* Patients with a history of neuromuscular disorders.

Ages: 20 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed at Mackay Memorial Hospital, the adult female patient was clinically assessed and diagnosed with urinary incontinence. Non-surgical treatments were administered, followed by subsequent monitoring and follow-up.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Urodynamic study (intravesical pressure) | form the baseline to the post-treatment measurement (about 6 month post)
  intravesical pressure (cmH2O)
Urodynamic study (abdominal pressure) | form the baseline to the post-treatment measurement (about 6 month post)
  abdominal pressure (cmH2O)
Urodynamic study (detrusor pressure) | from the baseline to the post-treatment measurement (about 6 month post)
  detrusor pressure (cmH2O)
Urodynamic study (Infused volume) | from the baseline to the post-treatment measurement (about 6 month post)
  infused volume (ml)
Urodynamic study (voided volume) | from the baseline to the post-treatment measurement (about 6 month post)
  voided volume (ml)
Pad test | from the baseline to the post-treatment measurement (about 6 month post)
  The weight of Pad (g) before and after testing
Bladder diary (voiding frequency) | from the baseline to the post-treatment measurement (about 6 month post)
  the daily voiding frequency (times)
Bladder diary (voiding volume) | from the baseline to the post-treatment measurement (about 6 month post)
  the daily voiding volume (ml)
Questionaire (UDI-6) | from the baseline to the post-treatment measurement (about 6 month post)
  The urogenital distress inventory-6 (UDI-6)
Questionaire (IIQ-7) | from the baseline to the post-treatment measurement (about 6 month post)
  incontinence impact questionnaire-7 (IIQ-7)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Hsuan Lau, M.D., Study Chair — Department of Ear, Nose, and Throat, MacKay Memorial Hospital, Taipei, Taiwan
Locations (1):
- Department of Obstetrics and Gynecology, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
For we uncertain if this might violate personal information laws in our country.

REFERENCES:
- [Background] Denisenko AA, Clark CB, D'Amico M, Murphy AM. Evaluation and management of female urinary incontinence. Can J Urol. 2021 Aug;28(S2):27-32. PMID 34453426
- [Background] Wallace SL, Miller LD, Mishra K. Pelvic floor physical therapy in the treatment of pelvic floor dysfunction in women. Curr Opin Obstet Gynecol. 2019 Dec;31(6):485-493. doi: 10.1097/GCO.0000000000000584. PMID 31609735
- [Background] Aoki Y, Brown HW, Brubaker L, Cornu JN, Daly JO, Cartwright R. Urinary incontinence in women. Nat Rev Dis Primers. 2017 Jul 6;3:17042. doi: 10.1038/nrdp.2017.42. PMID 28681849
- [Background] Lin HY, Tsai HW, Tsui KH, An YF, Lo CC, Lin ZH, Liou WS, Wang PH. The short-term outcome of laser in the management of female pelvic floor disorders: Focus on stress urine incontinence and sexual dysfunction. Taiwan J Obstet Gynecol. 2018 Dec;57(6):825-829. doi: 10.1016/j.tjog.2018.10.010. PMID 30545535
- [Derived] Lau HH, Lai CY, Hsieh MC, Peng HY, Chou D, Su TH, Lee JJ, Lin TB. Effect of intra-vaginal electric stimulation on bladder compliance in stress urinary incontinence patients: the involvement of autonomic tone. Front Neurosci. 2024 Aug 7;18:1432616. doi: 10.3389/fnins.2024.1432616. eCollection 2024. PMID 39170685